CLINICAL TRIAL: NCT04562285
Title: Initial and Sustained Immunity to SARS-CoV-2 Measured by Serologic Assays on an Automated Immunoassay System
Brief Title: Sustained Immunity to COVID-19 as Measured by SARS-CoV-2 Serology Assays
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Bernard Cook, Division Head, Chemistry-Pathology, Henry Ford Health System
Other Study IDs: 13978
Record Dates: First submitted 2020-09-22; First posted 2020-09-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Covid19
Keywords: SARS-CoV-2; Antibodies; Seroprevalence
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Serologic immunoassays to SARS-CoV-2 antibodies — Detect and characterize antibodies to SARS-CoV-2

SUMMARY:
The primary objective is to assess the ability of COVID-19 IgG and IgM assays to detect an immune response in COVID-19 patients in the Henry Ford Health System (HFHS), both during hospitalization and over the following 12 months.

DETAILED DESCRIPTION:
The design strategy for this study is to validate the detection of COVID-19 antibodies in subjects at HFHS who test positive with RT-PCR for SARS-CoV-2 using fully automated test systems already in the core automated laboratory at HFH. This is a study of the immune response and kidney health of subjects who have recovered from COVID-19 infection.

There are 4 aims:

Aim 1. Assess detection of COVID-19 antibodies in subjects before discharge from HFHS who tested positive with RT-PCR for SARS-CoV-2 using fully automated immunoassays.

Aim 2. Evaluate emergence of immunity over a one-year period in subjects who tested positive with RT-PCR for SARS-CoV-2 using a fully-automated immunoassays.

Aim 3. Monitor renal function and kidney health at 6 and 12- months post diagnosis with COVID-19.

Aim 4. Determine if SAR-COV-2 can be detected in the saliva of patients over a one year period after a positive PCR test.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age
* Positive COVID-19 by RT-PCR SARS-CoV-2 assay
* Patients must have a serum sample stored by pathology or within the TCRC biorepository around the date of their COVID-19 RT-PCR positive test

Exclusion Criteria:

* < 18 years of age
* negative for RT-PCR
* no serum sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects will be identified from a retrospective data review and a laboratory information system (LIS) SunQuest identification of COVID-19 positive (RT-PCR SARS CoV-2) samples or who are already participating in the TCRC collection protocol. This study will recruit subjects in which a baseline serum sample was already obtained either through standard of care procedures or through voluntary participation in the TCRC biorepository.
Sampling Method: Probability Sample
Enrollment: 829 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Detection of antibodies to SARS-CoV-2 in human serum and plasma | 12 months
  The study will assess the ability of COVID-19 IgG and IgM assays to detect an immune response in COVID-19 patients in the Henry Ford Health System (HFHS), both during hospitalization and over the following 12 months. The study will use Beckman Coulter anti-Spike IgG assay and Roche anti-Nucleocapsid assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No